CLINICAL TRIAL: NCT00424892
Title: A 6-Month Open-Label Extension Study of the Long-Term Safety of DVS SR in Outpatients With Fibromyalgia Syndrome.
Brief Title: Study Evaluating DVS SR in Patients With Fibromyalgia Syndrome
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3151A4-330
Record Dates: First submitted 2007-01-18; First posted 2007-01-22 (Estimated); Last update posted 2007-12-06 (Estimated); Status verified 2007-12

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

INTERVENTIONS:
Drug: Desvenlafaxine Sustained Release

SUMMARY:
The primary objective is to evaluate the long-term safety of desvenlafaxine succinate sustained-release (DVS SR) during open-label treatment in adult outpatients with fibromyalgia syndrome.

DETAILED DESCRIPTION:
Patients completing study 3151A4-327 have the opportunity to be treated with DVS SR during the 6 month extension study.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients who have completed double-blind treatment in study 3151A4-327 for fibromyalgia Syndrome with no major protocol violations and no events that would preclude the patient's entry into the long-term open-label study.
* Women of childbearing potential must have a negative serum pregnancy test result at study start.

Exclusion criteria:

* Presence of any new/and or clinically important medical condition that might compromise patient's safety.
* Use of prohibited treatment.
* Meets any of the exclusion criteria listed for study 3151A4-327.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600
Dates: Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
The following assessments are made to assess safety: physical examination, vital signs, standard 12-lead ECG, laboratory determinations, adverse events and serious adverse events, BDI-II.

SECONDARY OUTCOMES:
Pain score on the Numeric Rating Scale, FIQ score, PGIC, MAF, CGIC, Patient Global Symptom Rating and Physician Global Rating, MTPS, MOS-Sleep Measure.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (55):
- United States (55):
  - Huntsville, Alabama
  - Mobile, Alabama
  - Phoenix, Arizona
  - Anaheim, California
  - Sacramento, California
  - San Diego, California
  - Santa Ana, California
  - Walnut Creek, California
  - Denver, Colorado
  - Cromwell, Connecticut
  - Brooksville, Florida
  - DeLand, Florida
  - Delray Beach, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Palm Beach Gardens, Florida
  - Pembroke Pines, Florida
  - St. Petersburg, Florida
  - Sunrise, Florida
  - Tamarac, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Decatur, Georgia
  - Smyrna, Georgia
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Lexington, Kentucky
  - Rockville, Maryland
  - Boston, Massachusetts
  - Newton, Massachusetts
  - Lansing, Michigan
  - Kansas City, Missouri
  - St Louis, Missouri
  - Las Vegas, Nevada
  - Clementon, New Jersey
  - Raleigh, North Carolina
  - Cincinnati, Ohio
  - Dayton, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Duncansville, Pennsylvania
  - Harleysville, Pennsylvania
  - Philadelphia, Pennsylvania
  - Sellersville, Pennsylvania
  - West Reading, Pennsylvania
  - Warwick, Rhode Island
  - Charleston, South Carolina
  - Summerville, South Carolina
  - Bristol, Tennessee
  - Chattanooga, Tennessee
  - Memphis, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - San Antonio, Texas
  - Middleton, Wisconsin